CLINICAL TRIAL: NCT05915806
Title: Enteral Supplementation With High-dose Docosahexaenoic Acid on the Risk for Bronchopulmonary Dysplasia in Very Preterm Infants: A Collaborative Study Protocol for an Individual Participant Data Meta-analysis
Brief Title: Enteral High-dose DHA Supplementation on Bronchopulmonary Dysplasia in Very Preterm Infants: a Collaborative Study
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: CHU de Quebec-Universite Laval (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government); Laval University (Other); South Australian Health and Medical Research Institute (Other); McGill University Health Centre/Research Institute of the McGill University Health Centre (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MP-20-2015-2144; F1H-80784
Record Dates: First submitted 2023-05-30; First posted 2023-06-23 (Actual); Last update posted 2025-07-14 (Actual); Status verified 2025-07

CONDITIONS: Bronchopulmonary Dysplasia; Child Development; Neonatal and Perinatal Conditions
Keywords: Omega-3; Fatty acids; Preterm infants; Bronchopulmonary dysplasia; Individual participant data meta-analysis
MeSH Terms: conditions — Bronchopulmonary Dysplasia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The prior systematic review included a meta-analysis of aggregated data of trials that examined the effects of an enteral supplementation with high-dose DHA during the neonatal period on the risk for BPD (any definition), death, BPD severity (any definition) and a combined outcome of BPD or death in preterm infants born less than 29 weeks of gestation. Information on data sources (searched up to August 1st, 2022), search strategy, selection process, data extraction and risk of bias assessment were detailed in the prior protocol and publication. All four trials included in the prior systematic review will be considered for inclusion in this IPD meta-analysis.
  Upon the early period of selecting studies for the prior systematic review, the principal investigator (IM) has contacted the primary author of trials for potential agreement to share de-identified IPD for the purpose of this participant-level meta-analysis. All IPD datasets will be harmonised and combined into one large dataset.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- High-dose DHA (Experimental): Enteral supplementation with high-dose DHA in the neonatal period.
  Interventions: Dietary Supplement: High-dose DHA
- Control (Placebo Comparator): Control.
  Interventions: Dietary Supplement: Control

INTERVENTIONS:
Dietary Supplement: High-dose DHA — Direct enteral DHA supplementation at a dose of at least 40 mg/kg/day or DHA supplementation of breast milk or formula aiming for at least 0.4% of total fatty acids.
  Arms: High-dose DHA
Dietary Supplement: Control — Control with no or low-dose DHA.
  Arms: Control

SUMMARY:
This one-stage individual participant data (IPD) meta-analysis study will aim to determine whether high-dose docosahexaenoic acid (DHA) enteral supplementation during the neonatal period is associated with the risk for severe bronchopulmonary dysplasia (BPD) at 36 weeks' postmenstrual age (PMA) compared to control, in contemporary cohorts of preterm infants born at less than 29 weeks of gestation. The association between high-dose DHA and severe BPD will also be explored in important subgroups according to sex, gestational age, small-for-gestational age and mode of delivery.

DETAILED DESCRIPTION:
Severe BPD is a well-known factor consistently associated with impaired cognitive outcomes. Regarding reported benefits on long-term neurodevelopmental outcomes, the potential adverse effects of high-dose DHA supplementation on this short-term neonatal morbidity needs further investigations in infants born very preterm.

Therefore, based on previous systematic review findings and a known association between more severe BPD and unfavorable neurodevelopmental outcomes, a deeper understanding of the association between DHA and severe BPD needs further investigations. Harmonization of the severe BPD definition across the recent DHA trials, reclassified according to modern criteria will strengthen the results and allow their interpretation in balance with the potential efficacy of DHA on long-term neurodevelopmental outcomes. Moreover, inconsistent differential responses of DHA on BPD were previously reported according to subgroups such as sex, gestational age and mode of delivery and need to be further explored in this more vulnerable population.

ELIGIBILITY:
Trials included in our prior systematic review and traditional meta-analysis will be eligible for this IPD meta-analysis if they were registered randomized clinical trials of infants born preterm at less than 29 weeks of gestation and with adequate levels of blinding and allocation concealment. Moreover, eligibility will be restricted to trials conducted in a population of infants born after 2010 receiving contemporary respiratory care, similar to Jensen's cohort within which the severity-based definition of BPD was developed.

The intervention has to involve enteral administration of high-dose DHA supplementation during the neonatal period. A high-dose DHA supplementation is defined as direct enteral DHA supplementation at a dose of at least 40 mg/kg/day or DHA supplementation of breast milk or formula aiming for at least 0.4% of total fatty acids. The intervention should be randomly assigned as either enteral administration of high-dose DHA supplementation OR a control with no or low-dose DHA.

Trials evaluating intravenous DHA interventions or combined interventions (e.g. DHA combined to other nutrients or long-chain polyunsaturated fatty acids) are not considered for inclusion in this IPD meta-analysis to isolate the DHA effects and avoid heterogeneity in the intervention.

The IPD meta-analysis will be conducted using a harmonized severity-based definition of BPD in eligible trials. This definition will be based on Jensen's criteria that adequately predict childhood outcomes in a contemporary cohort of infants born very preterm. To be included, prospectively collected data from eligible trials should allow BPD severity outcome classification and harmonization according to Jensen's severity-based BPD criteria at 36 weeks' PMA.

Max Age: 14 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 1801 (Actual)
Dates: Start 2023-07-30 (Actual); Primary Completion 2023-11-15 (Actual); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Severe BPD | At 36 weeks' PMA
  A priori defined based on a team consensus, grades of severity (no BPD, grade 1-, 2-, 3-BPD) are defined on the mode of respiratory support at 36 weeks' PMA, regardless of prior or current oxygen therapy according to Jensen's criteria.
  Infants will be classified as severe BPD (Yes) if they presented a "grade 2- or 3-BPD" at 36 weeks' PMA, the two most severe grades of BPD according to Jensen's classification. Grade 2 is defined as respiratory support with nasal cannula >2 L/min ("high" flow) or noninvasive positive airway pressure (including nasal intermittent positive pressure ventilation or nasal continuous positive airway pressure). Grade 3 is defined as use of invasive mechanical ventilation.
  Infants will be classified as not severe BPD (No) if they presented "no BPD or grade 1-BPD" at 36 weeks' PMA. No BPD is defined as no support. Grade 1 is defined as respiratory support with nasal cannula ≤2 L/min ("low" flow).

SECONDARY OUTCOMES:
"Grade 2- or 3-BPD or death" | At 36 weeks' PMA
  Mortality is defined as death from any cause before 36 weeks' PMA and "Grade 2- or 3-BPD" is defined using Jensen's classification as previously described.
Severity grades of BPD | At 36 weeks' PMA
  Defined as no BPD, grade 1-, 2- or 3-BPD according to Jensen's criteria as previously described.
Mortality | Up to 36 weeks' PMA
  Defined as death from any cause.

OTHER OUTCOMES:
Rate of serious brain injury | Up to 40 weeks' PMA
  Defined as intraventricular hemorrhage of grade 3 or 4 or periventricular leukomalacia.
Rate of severe retinopathy of prematurity (ROP) | Up to 40 weeks' PMA
  Defined as unilateral or bilateral ROP of stages 4 or 5 or any stage of ROP requiring any treatment.
Neonatal morbidity count | Up to 40 weeks' PMA
  Including "grade 2- or 3-BPD", serious brain injury and severe ROP. A score from 0 to 3 will be attributed according to the presence or absence of each morbidity.
Rate of patent ductus arteriosus | Up to 40 weeks' PMA
  Defined as any patent ductus arteriosus requiring surgical treatment.
Rate of necrotising enterocolitis | Up to 40 weeks' PMA
  Defined as any necrotising enterocolitis requiring surgery.
Rate of culture-proven sepsis | Up to 40 weeks' PMA
  Defined as any episode of sepsis confirmed by positive blood culture and requiring antibiotics for therapeutic intent.
Child's weight | Up to 36 weeks' PMA
  Child anthropometry (i.e. weight in grams).
Child's length | Up to 36 weeks' PMA
  Child anthropometry (i.e. length in cm).
Child's head circumference | Up to 36 weeks' PMA
  Child anthropometry (i.e. head circumference in cm).

CONTACTS AND LOCATIONS:
Overall Officials: Isabelle Marc, MD, PhD, Principal Investigator — CHU de Québec-Université Laval; Pascal M. Lavoie, MD, PhD, Principal Investigator — University of British Columbia; Andrew J. McPhee, MB, BS, Principal Investigator — South Australian Health and Medical Research Institute; Carmel T. Collins, PhD, Principal Investigator — South Australian Health and Medical Research Institute; David Simonyan, MSc, Principal Investigator — CHU de Québec-Université Laval; Etienne Pronovost, BSc, Principal Investigator — CHU de Québec-Université Laval; Mireille Guillot, MD, Principal Investigator — CHU de Québec-Université Laval; Jacqueline F. Gould, PhD, Principal Investigator — South Australian Health and Medical Research Institute; Ibrahim Mohamed, MD, PhD, Principal Investigator — St. Justine's Hospital; Marc Beltempo, MD, Principal Investigator — McGill University Health Centre/Research Institute of the McGill University Health Centre; Amélie Boutin, PhD, Principal Investigator — CHU de Québec-Université Laval; Isabel Fortier, PhD, Principal Investigator — Research Institute of the McGill University Health Centre; Thomas R. Sullivan, PhD, Principal Investigator — South Australian Health and Medical Research Institute; Lynne Moore, PhD, Principal Investigator — Laval University; Maria Makrides, PhD, Principal Investigator — South Australian Health and Medical Research Institute
Locations (1):
- CHU de Québec-Université Laval, Québec, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No
There are currently no plan to share IPD obtained during this IPD meta-analysis. However, principal investigators will examine request from any groups for future collaboration.

REFERENCES:
- [Background] Marc I, Boutin A, Pronovost E, Guillot M, Bergeron F, Moore L, Makrides M. High doses of enteral docosahexaenoic acid omega-3 supplementation for prevention of bronchopulmonary dysplasia in very preterm infants: a protocol for a systematic review and meta-analysis. BMJ Open. 2022 Oct 17;12(10):e064515. doi: 10.1136/bmjopen-2022-064515. PMID 36253040
- [Background] Marc I, Boutin A, Pronovost E, Perez Herrera NM, Guillot M, Bergeron F, Moore L, Sullivan TR, Lavoie PM, Makrides M. Association Between Enteral Supplementation With High-Dose Docosahexaenoic Acid and Risk of Bronchopulmonary Dysplasia in Preterm Infants: A Systematic Review and Meta-analysis. JAMA Netw Open. 2023 Mar 1;6(3):e233934. doi: 10.1001/jamanetworkopen.2023.3934. PMID 36943265
- [Background] Jensen EA, Dysart K, Gantz MG, McDonald S, Bamat NA, Keszler M, Kirpalani H, Laughon MM, Poindexter BB, Duncan AF, Yoder BA, Eichenwald EC, DeMauro SB. The Diagnosis of Bronchopulmonary Dysplasia in Very Preterm Infants. An Evidence-based Approach. Am J Respir Crit Care Med. 2019 Sep 15;200(6):751-759. doi: 10.1164/rccm.201812-2348OC. PMID 30995069
- [Background] Papile LA, Burstein J, Burstein R, Koffler H. Incidence and evolution of subependymal and intraventricular hemorrhage: a study of infants with birth weights less than 1,500 gm. J Pediatr. 1978 Apr;92(4):529-34. doi: 10.1016/s0022-3476(78)80282-0. PMID 305471
- [Background] Schmidt B, Asztalos EV, Roberts RS, Robertson CM, Sauve RS, Whitfield MF; Trial of Indomethacin Prophylaxis in Preterms (TIPP) Investigators. Impact of bronchopulmonary dysplasia, brain injury, and severe retinopathy on the outcome of extremely low-birth-weight infants at 18 months: results from the trial of indomethacin prophylaxis in preterms. JAMA. 2003 Mar 5;289(9):1124-9. doi: 10.1001/jama.289.9.1124. PMID 12622582
- [Derived] Marc I, Lavoie PM, Sullivan TR, Pronovost E, Boutin A, Beltempo M, Guillot M, Gould JF, Simonyan D, McPhee AJ, Mohamed I, Moore L, Makrides M. High-dose docosahexaenoic acid for bronchopulmonary dysplasia severity in very preterm infants: a collaborative individual participant data meta-analysis. Am J Clin Nutr. 2025 Apr;121(4):826-834. doi: 10.1016/j.ajcnut.2025.01.004. Epub 2025 Feb 24. PMID 40180500
- [Derived] Marc I, Lavoie PM, McPhee AJ, Collins CT, Simonyan D, Pronovost E, Guillot M, Gould JF, Mohamed I, Beltempo M, Boutin A, Fortier I, Sullivan TR, Moore L, Makrides M. Enteral supplementation with high-dose docosahexaenoic acid on the risk of bronchopulmonary dysplasia in very preterm infants: a collaborative study protocol for an individual participant data meta-analysis. BMJ Open. 2023 Jul 30;13(7):e076223. doi: 10.1136/bmjopen-2023-076223. PMID 37518076